CLINICAL TRIAL: NCT07361848
Title: Randomized Controlled Trial Evaluating the Effects of Long-Hold Yielding Isometric Exercise on Pain, Function, Vascularity, and Mechanical Properties of the Patellar Tendon in Competitive Weightlifting Athletes
Brief Title: Long-Hold Yielding Isometric Exercise for Patellar Tendinopathy in Weightlifting Athletes
Acronym: QuantFlow
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jaime Almazán Polo, Assistant Professor of Physiotherapy and Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCM-JAP-QUANTFLOW-26
Record Dates: First submitted 2025-12-01; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Patellar Tendinopathy / Jumpers Knee
Keywords: patellar tendinopathy; long hold yielding isometrics; weightlifting athletes; tendon vascularity; shear-wave elastography; quantitative ultrasound; echotexture; echostructure; ehointensity; echovariation; doppler imaging; tendon stifness; stress-strain curve; young's modulus; biomechanics; jumper's knee; iPulley isokinetic; countermovement jump; force platform biomechanics; tissue mechanical properties; musculoskeletal imaging; clincal trial; randomized controlled trial

STUDY DESIGN:
Intervention Model Description: This study uses a two-arm parallel-group randomized controlled design. Participants are assigned in a 1:1 ratio to either the Long-Hold Yielding Isometric intervention group or the usual-care control group. Randomization is computer-generated with allocation concealment. Outcome assessors for ultrasound imaging, elastography, and biomechanical testing are blinded to group assignment. The intervention lasts 8 weeks, with additional follow-up assessments at 12 and 24 weeks to evaluate durability of effects. The model is designed to compare therapeutic and mechanobiological responses between groups while accounting for sex stratification to explore gender-related differences in tendon adaptation.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessors are masked to group allocation. Ultrasound technicians, elastography operators, and biomechanical evaluators remain blinded throughout all assessment time points (T0, T1, T2, T3). Due to the nature of the exercise-based intervention, neither participants nor care providers can be blinded. Investigators responsible for data analysis will work with anonymized, coded datasets to maintain allocation concealment during statistical procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-Hold Yielding Isometrics (Experimental): This arm receives a structured long-hold yielding isometric (LH-YI) exercise program targeting the patellar tendon. Participants perform 3-5 sets of 3-5 repetitions, each consisting of a 30-60 second sustained isometric contraction at a discomfort level of 3-4/10. Exercises are performed three times per week for 8 weeks, using a yielding squat or mid-range knee-flexion isometric position. Load is individualized based on tolerance. One supervised session per week ensures correct technique and monitoring. The protocol aims to improve pain, tendon vascularity, stiffness, and neuromechanical performance through prolonged tendon loading.
  Interventions: Behavioral: Long-Hold Yielding Isometric Exercise Program
- Usual-Care Training Condition (Active Comparator): This arm follows standard training recommendations for patellar tendinopathy without exposure to long-duration isometric loading. Participants maintain their regular weightlifting training with guidance on load management, symptom monitoring, and progressive strengthening. No sustained isometric exercises are permitted. This condition serves as a real-world comparable control to evaluate the specific effects of long-hold yielding isometrics on pain, function, tendon vascularity, stiffness, and neuromechanical performance.
  Interventions: Other: Usual-Care Training Condition

INTERVENTIONS:
Behavioral: Long-Hold Yielding Isometric Exercise Program — The intervention consists of a structured long-hold yielding isometric (LH-YI) loading program targeting the patellar tendon. Participants perform 3-5 sets of 3-5 repetitions, each held for 30-60 seconds at an intensity corresponding to 3-4/10 discomfort. Exercises are executed in a controlled knee-flexion position, either as a yielding squat or machine-assisted isometric hold. Training takes place three times per week for 8 weeks, with one supervised session weekly to ensure correct load, technique, adherence, and safety. The protocol aims to induce mechanotransductive adaptation, reduce pain, modulate tendon vascularity, and improve tendon stiffness and neuromechanical performance.
  Other Names: Long-Hold Isometric Loading
  Arms: Long-Hold Yielding Isometrics
Other: Usual-Care Training Condition — Participants maintain their regular weightlifting training following standard recommendations for patellar tendinopathy management. This includes load monitoring, symptom-guided progression, avoidance of high-irritability movements, and general strengthening. No long-duration isometric exercises or targeted LH-YI loading are permitted. This condition serves as an active comparator reflecting real-world practice to isolate the specific therapeutic and mechanobiological effects of the long-hold yielding isometric protocol.
  Other Names: Standard Tendinopathy Management
  Arms: Usual-Care Training Condition

SUMMARY:
The goal of this clinical trial is to evaluate whether a long-hold yielding isometric exercise program improves pain, tendon vascularity, mechanical properties, and functional performance in weightlifting athletes with patellar tendinopathy. The study will also explore the safety and feasibility of this exercise strategy.

Researchers will compare the long-hold isometric intervention with routine training recommendations to determine its effects on symptoms and tendon function.

Participants will perform the supervised isometric protocol and complete pain ratings, functional tests, and ultrasound evaluations of the patellar tendon.

DETAILED DESCRIPTION:
This randomized controlled trial is part of the QuantFlow research program, a multidisciplinary initiative designed to advance the understanding of patellar tendon pathology through the integration of quantitative ultrasound imaging, Doppler-based intratendinous vascularity assessment, shear-wave elastography, biomechanical performance testing, and clinical evaluation. Within this framework, the present trial evaluates the therapeutic, mechanobiological, and functional effects of a long-hold yielding isometric exercise protocol in competitive weightlifting athletes with vascularized patellar tendinopathy.

Patellar tendinopathy is a common overload-related condition in Olympic weightlifting due to the repetitive exposure to high mechanical loads during movements such as deep squats, cleans, jerks, and ballistic pulling actions. These demands can result in localized tendon pain, reduced load tolerance, and impaired athletic performance. Ultrasound imaging in symptomatic athletes frequently reveals increased tendon thickness, hypoechoic regions, altered fibrillar organization, and varying degrees of Doppler-detected intratendinous vascularity. Although the clinical relevance of vascularity remains debated, its presence may be associated with pain modulation and tissue remodeling. Understanding how targeted tendon-loading strategies influence vascularity, stiffness, structure, and symptoms is therefore central to this trial.

Long-hold yielding isometric loading is a specific exercise strategy characterized by sustained tendon loading for extended durations, typically lasting 30 to 60 seconds per repetition. Compared with short-duration isometric contractions, prolonged loading is thought to stimulate mechanotransductive pathways more effectively, potentially promoting collagen reorganization, modulation of tendon stiffness, and improvements in neuromuscular efficiency. Prolonged isometric loading may also induce short-term analgesic effects and influence intratendinous vascular responses. However, evidence supporting these mechanisms in high-performance weightlifting athletes is limited, and randomized controlled trials in this population are scarce.

The study follows a two-arm, parallel-group randomized controlled design with four assessment time points: baseline, post-intervention at 8 weeks, and follow-up assessments at 12 and 24 weeks. Participants are competitive weightlifting athletes aged 18 to 45 years who train at least three times per week and present with symptomatic patellar tendinopathy of at least six weeks' duration and a baseline VISA-P score below 80. Ultrasound confirmation of structural tendon changes or Doppler-detected vascularity is required. Key exclusion criteria include previous patellar tendon surgery, tendon rupture, recent injection therapies, systemic conditions affecting tendon health, significant concomitant knee pathology, pregnancy, or inability to comply with the study protocol.

Baseline assessments include pain evaluation during tendon-loading activities using the Numeric Pain Rating Scale, functional disability assessed with the VISA-P questionnaire, high-resolution B-mode ultrasound for tendon morphology, Doppler ultrasound for vascularity assessment, and shear-wave elastography for quantification of tendon stiffness. Neuromechanical performance is evaluated using force plate-based countermovement and reactive jump testing, providing measures such as jump height, force-time characteristics, impulse, and rate of force development. Maximal isometric force is assessed using standardized isometric testing procedures. All assessments follow standardized acquisition protocols to ensure reproducibility and inter-session reliability.

Participants are randomly allocated to either the intervention group or a usual-care control group using a computer-generated randomization schedule with allocation concealment. Outcome assessors for imaging and biomechanical testing are blinded to group assignment. The intervention group completes a long-hold yielding isometric exercise program consisting of three to five sets of three to five repetitions, each held for 30 to 60 seconds at a target discomfort level of 3 to 4 out of 10. Exercises are performed three times per week for eight weeks. The control group continues their usual training under standard tendinopathy management recommendations without exposure to long-duration isometric loading.

In addition to the primary and secondary outcome analyses, pre-specified exploratory subgroup analyses will be conducted stratified by biological sex (men and women) to examine whether sex modifies the response to the intervention. These analyses will be performed separately for key clinical, imaging, and biomechanical outcomes, including pain, functional status, tendon vascularity, tendon stiffness, and selected performance measures. The purpose of these analyses is exploratory and hypothesis-generating, and they are not intended to define additional independent outcome measures.

All primary and secondary outcome measures are reassessed at the post-intervention time point, with follow-up evaluations conducted at 12 and 24 weeks to determine the persistence of clinical, structural, and functional adaptations. Data quality is ensured through standardized operating procedures, routine quality-control checks, and secure data management practices. The study is conducted in accordance with international ethical standards for human research, including the principles of the Declaration of Helsinki and Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

1. Competitive weightlifting athletes (Olympic weightlifting or CrossFit) training ≥3 times per week.
2. Age 18-45 years.
3. Symptom duration of at least 6 weeks.
4. Presence of vascularized patellar tendinopathy, defined as Doppler-detectable intratendinous neovascularization using standardized settings.
5. VISA-P score < 80 at baseline.
6. Ability to perform loaded lower-limb exercises safely.
7. Willingness to refrain from other structured isometric interventions focused on the patellar tendon during the study period.
8. Ability to provide informed consent.
9. Sex/Gender requirement: both men and women eligible; the study includes sex-stratified analysis to examine potential sex-based differences in tendon response.

Exclusion Criteria:

1. Previous knee surgery within the past 12 months.
2. Partial or complete patellar tendon rupture (confirmed clinically or by ultrasound).
3. Coexisting knee conditions (e.g., meniscal tear, ACL/PCL injury, patellofemoral joint instability) that significantly affect load tolerance.
4. Systemic diseases affecting tendon health (e.g., diabetes, rheumatoid arthritis, connective tissue disorders).
5. Corticosteroid injection in the patellar tendon within the last 6 months.
6. Participation in other clinical trials involving exercise or tendon-loading interventions.
7. Neuromuscular or medical conditions limiting safe performance of isometric or plyometric exercise.
8. Pregnancy.
9. Inability to commit to follow-up assessments at 8, 12, and 24 weeks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2027-02-01 (Estimated); Primary Completion 2027-12-20 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Functional Disability (Victorian Institute of Sport Assessment Scale for Tendinopathy, VISA-P Score) | Baseline, 8 weeks (post-intervention), 12 weeks follow-up, 24 weeks follow up
  Patellar tendon-related functional impairment assessed using the Victorian Institute of Sport Assessment for Patellar Tendinopathy (VISA-P) questionnaire (0-100). Higher scores indicate better function. This measure evaluates global clinical improvement and load tolerance in daily living and sports context.
Pain During Tendon-Loading Activities (Numeric Pain Rating Scale) | Baseline, 8 weeks (post-intervention), 12 weeks follow-up, and 24 weeks follow-up
  Pain intensity during tendon-loading activities, such as squatting or jumping, assessed using the Numeric Pain Rating Scale (NPRS, 0-10), where 0 represents no pain and 10 represents the worst pain imaginable. Higher scores indicate greater pain. This outcome reflects symptom severity and clinical response to the intervention.
Patellar Tendon Vascularity (Surface Area Quantification) | Baseline and 8 weeks (post-intervention)
  Quantitative assessment of intratendinous vascularity using Surface Area Quantification (SAQ) derived from power Doppler ultrasound images. Doppler images are processed using image segmentation in Fiji/ImageJ software to isolate Doppler-positive pixels within a predefined tendon region of interest. Vascularity is expressed as the percentage of Doppler-positive pixel area relative to the total tendon area analyzed, with higher percentages indicating greater intratendinous vascularization.
Patellar Tendon Vascularity (Öhberg Score) | Baseline and 8 weeks (post-intervention)
  Intratendinous neovascularization assessed using the Öhberg grading scale based on power Doppler ultrasound imaging. The scale ranges from 0 to 4, where 0 indicates absence of Doppler-detected vessels and higher scores indicate increasing degrees of intratendinous neovascularization. Higher scores represent greater vascularity.
Patellar Tendon Vascularity (Modified Öhberg Score) | Baseline and 8 weeks (post-intervention)
  Intratendinous neovascularization assessed using the Modified Öhberg grading scale based on power Doppler ultrasound imaging. The scale ranges from 0 to 5, reflecting the proportion and extent of Doppler-detected intratendinous vessels within the region of interest, with higher scores indicating greater vascularity.
Tendon echostructure: Patellar Tendon Cross-Sectional Area (CSA) | Baseline, 8 weeks (post-intervention)
  Patellar tendon cross-sectional area (CSA, square millimeters [mm²]) will be assessed using transverse B-mode ultrasound imaging. CSA will be measured at three standardized locations along the tendon (proximal, mid-portion, and distal), and the mean value across the three regions will be calculated and used for analysis. CSA reflects tendon morphology and structural adaptation to mechanical loading.
Tendon echostructure: Patellar Tendon Thickness | Baseline, 8 weeks (post-intervention)
  Patellar tendon thickness (millimeters [mm]) will be measured using longitudinal B-mode ultrasound imaging at three standardized locations along the tendon (proximal, mid-portion, and distal). The mean thickness across the three regions will be calculated and used for analysis. Tendon thickness represents a structural characteristic associated with tendon adaptation and pathological changes.

SECONDARY OUTCOMES:
Tendon Stiffness (Shear-Wave Elastography in kPa) | Baseline, 8 weeks (post-intervention)
  Patellar tendon mechanical stiffness quantified using shear-wave elastography and expressed in kilopascals (kPa). Shear-wave elastography provides a continuous quantitative measure of tissue shear modulus, with higher kPa values indicating greater tendon stiffness. Three repeated elastography measurements will be obtained at each assessment and averaged for analysis. Changes in tendon stiffness will be evaluated by comparing values across assessment time points.
Tendon Stiffness (Shear-Wave Velocity) | Baseline and 8 weeks (post-intervention)
  Patellar tendon mechanical stiffness quantified using shear-wave elastography and expressed as shear-wave propagation velocity in meters per second (m/s). Shear-wave velocity provides a continuous quantitative measure of tissue stiffness, with higher velocity values indicating greater tendon stiffness. Three repeated elastography measurements will be obtained at each assessment and averaged for analysis. Changes in tendon stiffness will be evaluated by comparing values across assessment time points.
Tendon Mechanical Properties: Stiffness (iPulley and Ultrasound) | Baseline, 8 weeks (post-intervention)
  Patellar tendon mechanical stiffness in newtons per millimeter (N/mm) will be quantified using synchronized force and ultrasound-based tendon elongation measurements obtained during isometric loading tasks. Tendon force-elongation curves will be generated, and stiffness will be calculated as the slope of the linear regression between tendon force and tendon elongation within the linear region of the loading curve, defined between 50% and 100% of the maximal tendon force. Higher stiffness values indicate greater resistance of the tendon to deformation under tensile load.
Maximal Isometric Force (IMTP or iPulley) | Baseline, 8 weeks (post-intervention)
  Peak isometric force and force-time characteristics measured using an isometric mid-thigh pull setup (TrueStrenght, Hawkins Dynamics) or the iPulley system.
Tendon Echointensity (B-mode Ultrasound, Echotexture) | Baseline, 8 weeks (post-intervention)
  Quantitative echointensity of the patellar tendon assessed from standardized B mode ultrasound images. Echointensity is defined as mean grayscale pixel brightness within a standardized region of interest (ROI), reflecting collagen organization and tissue integrity.
Tendon Echovariation (B-mode Ultrasound, Echotexture) | Baseline and 8 weeks (post-intervention)
  Quantitative echovariation of the patellar tendon assessed from standardized B-mode ultrasound images. Echovariation is defined as the coefficient of variation of grayscale pixel intensities within a standardized region of interest (ROI), calculated as:
  Echovariation (%) = (standard deviation of pixel intensities / mean echointensity) × 100 This metric represents grayscale texture heterogeneity and microstructural irregularity commonly associated with tendinopathic changes.
Plyometric Performance Metrics: Reactive Strength Index (Force Plate Assessment) | Baseline and 8 weeks (post-intervention)
  Plyometric variables reflect neuromuscular efficiency, elastic energy utilization, and tendon-muscle unit performance relevant to competitive weightlifting athletes. Variables will be quantified using bilateral force plates during countermovement and reactive jump tasks.
  Reactive Strength Index (RSI) calculated as jump height divided by ground contact time during. RSI is reported as a dimensionless ratio.
Plyometric Performance Metrics: Jump Height (Force Plate Assessment) | Baseline, 8 weeks (post-intervention)
  Plyometric variables reflect neuromuscular efficiency, elastic energy utilization, and tendon-muscle unit performance relevant to competitive weightlifting athletes. Variables will be quantified using bilateral force plates during countermovement and reactive jump tasks.
  Jump Height, derived from impulse-momentum or flight-time methods obtained from force plate data. Jump height is expressed in centimeters (cm).
Plyometric Performance Metrics: Ground Contact Time (Force Plate Assessment) | Baseline and 8 weeks (post-intervention)
  Plyometric variables reflect neuromuscular efficiency, elastic energy utilization, and tendon-muscle unit performance relevant to competitive weightlifting athletes. Variables will be quantified using bilateral force plates during countermovement and reactive jump tasks.
  Ground contact time, defined as the duration of foot contact with the force platform prior to takeoff during reactive jump tasks. Ground contact time is expressed in milliseconds (ms).
Plyometric Performance Metrics: Flight time (Force Plate Assessment) | Baseline and 8 weeks (post-intervention)
  Plyometric variables reflect neuromuscular efficiency, elastic energy utilization, and tendon-muscle unit performance relevant to competitive weightlifting athletes. Variables will be quantified using bilateral force plates during countermovement and reactive jump tasks.
  Flight time, defined as the period during which vertical ground reaction force equals zero during the jump. Flight time is expressed in milliseconds (ms).
Tendon Mechanical Properties: Strain (iPulley and Ultrasound) | Baseline, 8 weeks (post-intervention)
  Maximum patellar tendon strain in percentage (%) will be calculated as the ratio between maximal tendon elongation measured during isometric loading and resting tendon length assessed at a standardized joint position. Tendon strain represents the relative deformation of the tendon under load and reflects tendon extensibility during force production.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Faculty of Nursing, Physiotherapy and Podiatry, Department of Physiotherapy, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) derived from this study may be shared after completion of the primary analyses and publication of the main results. Shared data will be limited to curated and filtered analytical datasets containing derived quantitative variables used in statistical analyses, such as ultrasound-derived morphology, vascularity and elastography metrics, biomechanical outcomes, and clinical scale scores. Raw data sources, including original imaging files, force recordings and questionnaire forms, will not be shared.
  All shared datasets will be fully anonymized in compliance with GDPR (EU 2016/679), Spanish LOPDGDD regulations and institutional ethical requirements. Access to de-identified IPD will be provided upon reasonable request, subject to review by the study investigators, and shared through secure institutional or trusted research repositories after publication of the primary study findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified individual participant data and supporting documents will be made available after publication of the primary study results. Data will remain available for a minimum of five years following initial release.
Access Criteria: Access to de-identified individual participant data and supporting information will be granted upon reasonable request for research purposes. Requests will be reviewed by the study investigators to assess scientific validity, ethical compliance and alignment with participant consent. Approved requests will receive access to curated and filtered analytical datasets only. Raw data sources, including imaging files and original questionnaires, will not be shared.
URL: https://biblioguias.ucm.es/docta/datosdeinvestigacion

REFERENCES:
- [Background] Pringels L, Van Acker G, Wezenbeek E, Burssens A, Vanden Bossche L. Novel Insights Into the Intratendinous Pressure Behavior of the Achilles Tendon in Athletes. Sports Health. 2025 Mar;17(2):374-382. doi: 10.1177/19417381241245357. Epub 2024 Apr 12. PMID 38610105
- [Background] Scattone Silva R, Song KE, Hullfish TJ, Sprague A, Silbernagel KG, Baxter JR. Patellar Tendon Load Progression during Rehabilitation Exercises: Implications for the Treatment of Patellar Tendon Injuries. Med Sci Sports Exerc. 2024 Mar 1;56(3):545-552. doi: 10.1249/MSS.0000000000003323. Epub 2023 Oct 16. PMID 37847102
- [Background] Merkel, M. F. R., Hellsten, Y., Magnusson, S. P., and Kjaer, M. 2021. Tendon blood flow, angiogenesis, and tendinopathy pathogenesis. Transl Sports Med 4:756-771. https://doi.org/10.1002/TSM2.280.